CLINICAL TRIAL: NCT06865430
Title: Management of Dysuria and Irritative Symptoms After HoLEP: a Prospective Study Evaluating the Efficacy of Alpha-Blocker Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ali Kaan Yildiz, principle investigator, Ankara Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: AŞH.AKYILDIZ.008
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Prostate Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GROUP USING ALPHA BLOCKERS (Active Comparator): Alpha blockers will be started and irritative symptoms will be questioned.
  Interventions: Drug: Tamsulosin Hydrochloride
- GROUP NOT USING ALPHA BLOCKERS (Placebo Comparator): Patients who were not started on alpha blockers will constitute this group.
  Interventions: Other: Sham

INTERVENTIONS:
Drug: Tamsulosin Hydrochloride — Alpha blockers will be started and symptoms will be questioned.
  Arms: GROUP USING ALPHA BLOCKERS
Other: Sham — Patients who were not started on alpha blockers will constitute this group.
  Arms: GROUP NOT USING ALPHA BLOCKERS

SUMMARY:
Holmium Laser Enucleation of the Prostate (HoLEP) is an increasingly popular endoscopic minimally invasive surgical technique for the treatment of benign prostatic hyperplasia (BPH). In the literature, the long-term efficacy and low complication rates of HoLEP have been highlighted in many studies. However, in the early postoperative period, particularly within the first three months, irritative symptoms are reported in 17-35% of cases (1-2).

The pathophysiology of postoperative irritative symptoms is not yet fully understood, but it has been suggested that these symptoms may be associated with urethral trauma, the mucosal healing process, and detrusor overactivity. These symptoms can significantly impact quality of life, reducing patient satisfaction. In particular, dysuria is a frequently encountered symptom after HoLEP, with considerable individual variability in its severity and duration.

The effectiveness of alpha-blockers in alleviating postoperative dysuria and irritative symptoms remains a topic of debate in the literature. Although prostate tissue is surgically removed, alpha-blockers may improve urinary flow and relieve symptoms associated with bladder outlet obstruction by reducing urethral smooth muscle tone (3). Studies on the use of alpha-blockers following transurethral resection of the prostate (TURP) have shown limited postoperative benefits (4). However, to the best of our knowledge, no study has specifically evaluated their use following HoLEP, an enucleation-based technique. Therefore, further studies are needed to assess the role of alpha-blockers in managing dysuria after HoLEP.

The aim of this study is to evaluate the effectiveness of alpha-blocker therapy in managing dysuria and other irritative symptoms following HoLEP. Additionally, the study seeks to determine the impact of this treatment on quality of life and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

Men over 40 years old, under 85 years old, and HoLEP surgery

Exclusion Criteria:

Prostate cancer, patients with bladder stones, patients with a history of urethral stricture, patients with detrusor underactivity in urodynamics, those who have had prostate surgery before

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-09-04 (Estimated); Study Completion 2026-03-04 (Estimated)

PRIMARY OUTCOMES:
dysuria vas score out of 10 points | ONE MONTH
urgency vas score out of 10 points | ONE MONTH
ıpps score | ONE MONTH

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara bilkent city hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No